CLINICAL TRIAL: NCT02528929
Title: Assessing the Clinical Response to a Gluten Free Diet in Patients With Diarrhoea Predominant Irritable Bowel Syndrome, in Whom Overt Coeliac Disease Has Been Excluded
Brief Title: Gluten-free Diet in Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STH16497
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Diet, Gluten-Free

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- At-risk serology (Active Comparator): Gluten-free diet
  Interventions: Dietary Supplement: Gluten-free diet
- Not at-risk serology (Active Comparator): Gluten-free diet
  Interventions: Dietary Supplement: Gluten-free diet

INTERVENTIONS:
Dietary Supplement: Gluten-free diet — Patients with IBS-D will commence a gluten-free diet for 6 weeks following dietetic input. They will be informed they do not have coeliac disease. They will however be blinded to whether or not they have any markers of at-risk serology. They will self-complete validated questionnaires over 6 weeks. Any subjects who opt to continue with a gluten-free diet thereafter of their own volition will be kept under observation as per routine clinical care.

SUMMARY:
To evaluate the effects of a gluten-free diet in irritable bowel syndrome.

DETAILED DESCRIPTION:
Irritable bowel syndrome with diarrhoea (IBS-D) is commonly encountered in primary and secondary-care practice. There are various triggers including diet. There is a growing number of people taking a gluten-free diet (GFD) of their own volition even in the absence of coeliac disease (CD). The investigators aim to assess whether a GFD could be of benefit to patients with IBS-D, previously naive to the effects of gluten and in whom CD has been excluded as per normal duodenal biopsies. The investigators will also assess whether certain factors may predict a clinical responder such as the presence or absence of at-risk coeliac serology.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 16 years or over
2. Patients fulfilling ROME III symptom based criteria for IBS-D but do not have coeliac disease

Exclusion Criteria:

1. Patients diagnosed with coeliac disease
2. Patients already on a gluten-free diet
3. Patients initially referred with self-reported gluten sensitivity
4. Patients with organic conditions that can mimic IBS-D such as idiopathic bile acid diarrhoea, pancreatic insufficiency, microscopic colitis, and inflammatory bowel disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-09; Primary Completion 2018-07-31 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome Symptom Severity Scores. This validated questionaire will be self-completed at baseline and at week 6. The investigators will compare the changes in scores over this time point. | 6 weeks

SECONDARY OUTCOMES:
Hospital Anxiety and Depression scores. This validated questionaire will be self-completed at baseline and at week 6. The investigators will compare the changes in scores over this time point. | 6 weeks
Fatigue Impact Scores. This validated questionaire will be self-completed at baseline and at week 6. The investigators will compare the changes in scores over this time point. | 6 weeks
Short-form 36 Quality of Life Scores. This validated questionaire will be self-completed at baseline and at week 6. The investigators will compare the changes in scores over this time point. | 6 weeks
Assess whether patients opt to continue with a GFD of their own volition | 1-2 years
  At the end of the six-week GFD trial period, patients will be asked whether or not they plan to continue with a GFD of their own volition. This will be assessed by a "yes/no" answer. Those who choose to do so will now be followed-up under routine clinical care over the next 1-2 years. This will allow the investigators to assess whether symptom-remission is maintained by using the same questionnaires mentioned in outcomes 1 to 4. It will also allow the investigators to monitor well-being in the form of body-mass index and serum haematinics (vitamin B12, folate, ferritin, albumin, haemoglobin).

CONTACTS AND LOCATIONS:
Overall Officials: David Sanders, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust

REFERENCES:
- [Derived] Aziz I, Trott N, Briggs R, North JR, Hadjivassiliou M, Sanders DS. Efficacy of a Gluten-Free Diet in Subjects With Irritable Bowel Syndrome-Diarrhea Unaware of Their HLA-DQ2/8 Genotype. Clin Gastroenterol Hepatol. 2016 May;14(5):696-703.e1. doi: 10.1016/j.cgh.2015.12.031. Epub 2015 Dec 31. PMID 26748221